CLINICAL TRIAL: NCT04307797
Title: A Pilot Study on the Effect of Glucagon and Glucagon-like Peptide-1 Co-agonism on Cardiac Function and Metabolism in Overweight Participants with Type 2 Diabetes (COCONUT)
Brief Title: Effect of Glucagon and Glucagon-like Peptide-1 Co-agonism on Cardiac Function and Metabolism in Overweight Participants with Type 2 Diabetes
Acronym: COCONUT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Antaros Medical (Industry)
Responsible Party: Principal Investigator, Dr Ian B Wilkinson, Professor of Therapeutics, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: COCONUT
Record Dates: First submitted 2020-02-19; First posted 2020-03-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Sodium Chloride; Exenatide; Maintenance; Glucagon

STUDY DESIGN:
Intervention Model Description: Single-centre, single-blinded, physiological pilot study
Who Masked: Participant
Masking Description: Imaging analysis performed by Antaros Medical (blinded to infusion)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: 0.9% Sodium-chloride — Part A - 0.9% saline infusion during cardiac PET-MRI scan
Drug: Exenatide (50ng/min for 30 minutes loading followed by 25ng/min maintenance) and glucagon 12.5ng/kg/min — Part A - exenatide and glucagon infusion during cardiac PET-MRI scan
  Other Names: Byetta
Drug: Glucagon 12.5ng/kg/min and 0.9% saline — Part A - Glucagon and 0.9% saline infusion during PET-MRI scan
Drug: 0.9% Sodium-chloride — Part B - 0.9% saline infusion during 7T 31P MRS scan
Drug: Exenatide (50ng/min for 30 minutes loading followed by 25ng/min maintenance) and glucagon 12.5ng/kg/min — Part B - exenatide and glucagon infusion during 7T 31P MRS scan
Drug: Glucagon 12.5ng/kg/min — Part B - Glucagon infusion during 7T 31P MRS scan

SUMMARY:
The study seeks to explore the cardiovascular effects of co-agonism at the glucagon and (glucagon-like peptide-1) GLP-1 receptor. Glucagon and exenatide will be intravenously infused into participants with type 2 diabetes (T2DM). Overall, the aim of the study is to further the investigator's understanding on the role these endogenous substances have on normal cardiac physiology, myocardial energetics and myocardial glucose uptake through a series of PET and MRI imaging studies

DETAILED DESCRIPTION:
This is a single-centre, single-blinded pilot study designed to understand the role the GLP-1 receptor agonist, exenatide, and glucagon receptor co-agonism has on normal cardiac physiology, myocardial energetics and myocardial glucose utilisation.

Part A - Overweight participants with type 2 diabetes will act as their own control and will undergo a series of three imaging studies (in a randomised order) as detailed below:

1. Cardiac positron emission tomography-magnetic resonance imaging (PET-MRI) with fluorine-18-fluorodeoxyglucose (18F-FDG) with placebo (0.9% saline) infusion
2. Cardiac PET-MRI with 18F-FDG with co-infusion of exenatide and glucagon
3. Cardiac PET-MRI with 18F-FDG with infusion of glucagon

Part B - Overweight participants with type 2 diabetes will act as their own control and will undergo a series of two imaging studies (in a randomised order), followed by one optional visit as detailed below:

1. 7T Phosphorus (P) 31 magnetic resonance spectroscopy (MRS) (31P-MRS) with placebo (0.9% saline) infusion
2. 7T 31P-MRS with co-infusion of glucagon and exenatide 3 (optional) 7T 31P-MRS with infusion of glucagon

Study outcome measures are detailed below

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate
* Aged >18 years
* Clinical diagnosis of T2DM, either diet controlled or treated with metformin (to be withheld on the morning of the imaging visit)
* BMI ≥25kg/m2
* Current non-smoker

Exclusion Criteria:

* Females of childbearing potential (Part A only) / current pregnancy (all parts)
* Sustained Hypertension (sustained BP >160/100mmHg) or hypotension (systolic BP below 90 mmHg)
* Clinically significant heart disease
* Implanted heart pacemaker or implantable cardioverter defibrillator (ICD)
* Known active malignancy other than skin cancer
* Known renal failure (creatinine >150µmol/L)
* Known type one diabetes mellitus / known or clinically suspected diagnosis of a monogenic form of diabetes
* Poorly controlled blood glucose
* Current daily use of anti-diabetic medication including Insulin, GLP-1 based agonists, DPP4i or any other medication known to interact with either of the study drugs (exenatide or glucagon)
* Current involvement in the active treatment phase of other research studies, (excluding observational/non-interventional).
* Contraindication for MRI/PET scan, i.e. any reason which precludes MRI imaging according to local policy (ie internal pacemaker/defibrillator, metal fragments, claustrophobia)
* Participation in research studies in the last 3 years involving radiation (if the effective dose exceeded 10mSv). This does not include any diagnostic or therapeutic exposures which were clinically justified.
* Any other clinical reason which may preclude entry in the opinion of the investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Part A - Myocardial glucose uptake | Comparison between scans over a maximum period of 16 weeks
  Difference in myocardial glucose uptake between 0.9% saline, glucagon:exenatide and glucagon scan as measured by 18F-FDG
Part A - Global longitudinal strain / global circumferential strain / global radial strain | Comparison between scans over a maximum period of 16 weeks
  Difference in global longitudinal strain / global circumferential strain / global radial strain between 0.9% saline, glucagon:exenatide and glucagon scan as measured by CMR
Part A - Ejection fraction | Comparison between scans over a maximum period of 16 weeks
  Difference in ejection fraction between 0.9% saline, glucagon:exenatide and glucagon scan as measured by CMR
Part A - Stroke volume | Comparison between scans over a maximum period of 16 weeks
  Difference in stroke volume between 0.9% saline, glucagon:exenatide and glucagon scan as measured by CMR
Part A - Cardiac output | Comparison between scans over a maximum period of 16 weeks
  Difference in cardiac output between 0.9% saline, glucagon:exenatide and glucagon scan as measured by CMR
Part B - Changes in phosphocreatine/adenosine (PCr/ATP) radio | Comparison between scans over a maximum period of 16 weeks
  Changes in PCr/ATP radio between 0.9% saline, glucagon:exenatide and glucagon (optional) in the mid-interventricular septum as a measure of cardiac energy status as measured by 7T phosphorus (P) 31 magnetic resonance spectroscopy (MRS)
Part B - Changes in absolute concentrations of PCr and ATP defined by AHA 17- segment territory as a measure of cardiac energy status (determined by 31P-MRS) | Comparison between scans over a maximum period of 16 weeks
  Changes in absolute concentrations of PCr and ATP between 0.9% saline, glucagon:exenatide and glucagon (optional) as defined by AHA 17-segment territory as a measure of cardiac energy status (determined by 7T 31P-MRS)

SECONDARY OUTCOMES:
Part A - End systolic/diastolic ventricular/atrial volumes | Comparison between scans over a maximum period of 16 weeks
  Difference in end systolic/diastolic ventricular/atrial volumes between 0.9% saline, glucagon:exenatide and glucagon scan as measured by CMR
Part A - Radial strain | Comparison between scans over a maximum period of 16 weeks
  Difference in radial strain between 0.9% saline, glucagon:exenatide and glucagon scan as measured by CMR
Part A - Global systolic/diastolic longitudinal/circumferential/radial strain rate | Comparison between scans over a maximum period of 16 weeks
  Difference in global systolic/diastolic longitudinal/circumferential/radial strain rate between 0.9% saline, glucagon:exenatide and glucagon scan as measured by CMR
Part A - Relationship between early and late filling (from mitral flow) | Comparison between scans over a maximum period of 16 weeks
  Difference in early and late filling (from mitral flow) between 0.9% saline, glucagon:exenatide and glucagon scan as measured by CMR
Part A/B - Heart rate | Comparison between infusions (placebo vs drug) over a maximum period of 16 weeks
  Difference in heart rate between 0.9% saline, glucagon:exenatide and glucagon
Part A/B - Blood pressure | Comparison between infusions (placebo vs drug) over a maximum period of 16 weeks
  Difference in blood pressure between 0.9% saline, glucagon:exenatide and glucagon
Part A/B - Glucose | Comparison between infusions (placebo vs drug) over a maximum period of 16 weeks
  Difference in glucose between 0.9% saline, glucagon:exenatide and glucagon
Part A/B - Glucagon | Comparison between infusions (placebo vs drug) over a maximum period of 16 weeks
  Difference in glucagon between 0.9% saline, glucagon:exenatide and glucagon
Part A/B - Insulin | Comparison between infusions (placebo vs drug) over a maximum period of 16 weeks
  Difference in insulin between 0.9% saline, glucagon:exenatide and glucagon
Part A/B - C-peptide | Comparison between infusions (placebo vs drug) over a maximum period of 16 weeks
  Difference in C-peptide between 0.9% saline, glucagon:exenatide and glucagon
Part A/B - fatty acids | Comparison between infusions (placebo vs drug) over a maximum period of 16 weeks
  Difference in fatty acids between 0.9% saline, glucagon:exenatide and glucagon
Part A/B - exenatide | Comparison between infusions (placebo vs drug) over a maximum period of 16 weeks
  Difference in exenatide between 0.9% saline, glucagon:exenatide and glucagon
Part A/B - Total GLP-1 and total active GLP-1 | Comparison between infusions (placebo vs drug) over a maximum period of 16 weeks
  Difference in GLP-1 between 0.9% saline, glucagon:exenatide and glucagon
Part A/B - gastric inhibitory polypeptide | Comparison between infusions (placebo vs drug) over a maximum period of 16 weeks
  Difference in gastric inhibitory polypeptide between 0.9% saline, glucagon:exenatide and glucagon

CONTACTS AND LOCATIONS:
Overall Officials: Ian Wilkinson, MD, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust and The University of Cambridge, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No